CLINICAL TRIAL: NCT06700681
Title: Safety and Efficacy of Remimazolam Compared With Propofol Under EEG DSA Guiding During Cardiac Electrophysiology Studies and Ablation: Randomized Controlled Trial
Brief Title: RCT Comparing Remimazolam With Propofol Under EEG DSA Guidance During Cardiac Electrophysiology Studies and Ablation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-06-005B
Record Dates: First submitted 2024-09-10; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Hemodynamic; Remimazolam; Propofol; Cardiac Electrophysiology
MeSH Terms: interventions — Propofol; remimazolam; Intubation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- TIVA with Propofol and intubation (Placebo Comparator): Patient received cardiac electrophysiology studies and ablation under TIVA with Propofol induction and maintenance and airway is maintained with intubation and controlled ventilation.
  Interventions: Drug: Propofol; Device: With intubation and controlled ventilation to maintain airway
- TIVA with Remimazolam and intubation (Experimental): Patient received cardiac electrophysiology studies and ablation under TIVA with Remimazolam induction and maintenance and airway is maintained with intubation and controlled ventilation.
  Interventions: Drug: Remimazolam; Device: With intubation and controlled ventilation to maintain airway
- TIVA with Propofol and non-Intubated (Experimental): Patient received cardiac electrophysiology studies and ablation under TIVA with Propofol induction and maintenance and airway is maintained with spontaneous ventilation without intubation(non-intubated).
  Interventions: Drug: Propofol; Device: Maintain spontaneous ventilation without intubation
- TIVA with Remimazolam and non-Intubated (Experimental): Patient received cardiac electrophysiology studies and ablation under TIVA with Remimazolam induction and maintenance and airway is maintained with spontaneous ventilation without intubation(non-intubated).
  Interventions: Drug: Remimazolam; Device: Maintain spontaneous ventilation without intubation

INTERVENTIONS:
Drug: Propofol — TIVA induction and maintain with Propofol.
  Arms: TIVA with Propofol and intubation; TIVA with Propofol and non-Intubated
Drug: Remimazolam — TIVA induction and maintain with Remimazolam.
  Arms: TIVA with Remimazolam and intubation; TIVA with Remimazolam and non-Intubated
Device: With intubation and controlled ventilation to maintain airway — Patient receives intubation and controlled ventilation to maintain airway.
  Arms: TIVA with Propofol and intubation; TIVA with Remimazolam and intubation
Device: Maintain spontaneous ventilation without intubation — Patient maintains spontaneous ventilation without intubation.
  Arms: TIVA with Propofol and non-Intubated; TIVA with Remimazolam and non-Intubated

SUMMARY:
Brief Summary:

The goal of this RCT is to compare the Safety and efficacy of remimazolam compared with propofol under EEG DSA guiding during cardiac electrophysiology studies and ablation. The main questions it aims to answer are:

* Is Remimazolam as efficacy as propofol in cardiac electrophysiology studies and ablation?
* Is Remimazolam lower hypotension episodes or lower vasopressor dosages compare with propofol in cardiac electrophysiology studies and ablation? If there is a comparison group: Researchers will compare [arm information] to see if [insert effects].

Researchers will compare Remimazolam to Propofol to see if Remimazolam is more feasible in cardiac electrophysiology studies and ablation.

Participants will receive either Remimazolam or Propofol sedation during study period.

ELIGIBILITY:
Inclusion Criteria:

* Patient receives scheduled cardiac electrophysiology studies and ablation by the same cardiologist(one of the study investigator).

Exclusion Criteria:

* With existing vasopressor or shock status
* Patient refusal or cannot finish Mini-Cog or QoR-15 preoperatively
* Canceled by cardiologist
* Allergy history to the anesthetics used in this study
* History of abnormal lung function or required oxygen therapy preoperative

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic stability--Vasopressor dosage | Introperative
  Total dosage of vasopressor used during the procedure

SECONDARY OUTCOMES:
Respiratory depression require intubation | Introperative
  The incidence of patients in non-intubated groups receive intubation
TIVA failure rate | Introperative
  The incidence of TIVA shift to inhalation anesthetics
LOC time | Introperative
  Time from start induction to loss of conscious
Emergence time | Introperative
  Time from stop intravenous anesthetics infusion to eye opening
Sanctification of cardiologist | Perioperative
  The sanctification score of the cardiologist
QoR-15 | Preoperative to post-operative day 1
  The result of QoR-15 score
Mini-Cog | Preoperative to post-operative day 1
  The result of Mini-Cog score
Length of hospital stay | Upto 1 month
  Length of hospital stay
Adverse outcome | Upto 1 month
  Any adverse outcome
Length of CU stay | Upto 1 month
  Length of CU stay

CONTACTS AND LOCATIONS:
Overall Officials: Li Yi-Shiuan, Bachelor's, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No